CLINICAL TRIAL: NCT05939297
Title: The Turkish Adaptation, Validity and Reliability of the Heart Health Self-Efficacy and Self-Management Scale
Brief Title: Turkish Adaptation of Heart Health Self-efficacy and Self-Management Scale
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Tunç Süygün, LECTURER, Karamanoğlu Mehmetbey University
Other Study IDs: KMU-TUNCSUYGUN-002
Record Dates: First submitted 2023-06-21; First posted 2023-07-11 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; validitiy; reliability; Self efficacy; Self Management; Heart Health
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- people with coronary heart disease: In order to measure the self-management and self-efficacy levels of the patients,Heart Health Self-efficacy and Self-Management Scale , Self-Care Management Scale in Chronic Diseases, general self-efficacy scales will be applied to the patients.
  Interventions: Other: Heart Health Self-efficacy and Self-Management Scale; Other: Self-Care Management Scale in chronic diseases; Other: general self-efficacy scale

INTERVENTIONS:
Other: Heart Health Self-efficacy and Self-Management Scale — In order to measure the self-management and self-efficacy levels of the individuals, patients will be administered the Heart Health Self-efficacy and Self-Management Scale.
Other: Self-Care Management Scale in chronic diseases — For the external construct validity statistical method, the self-management level of the individuals will also be determined with the Self-Care Management in Chronic Diseases Scale, which has been previously validated and reliable in Turkish.
Other: general self-efficacy scale — For the external construct validity statistical method, the self-efficacy level of the individuals will also be determined with the general self-efficacy scale, which has been previously validated and reliable in Turkish.

SUMMARY:
The importance of lifestyle changes to control risk factors in the prevention, treatment and management of coronary heart disease (CHD), a major health problem, has been emphasised. In addition, physical, social, psychological and occupational limitations arising from the disease negatively affect the quality of life and self-efficacy perceptions of individuals, making it difficult to comply with treatment and disease management. There are general self-efficacy and self-management scales for which Turkish validity and reliability studies have been conducted previously. However, these scales are not specific to coronary heart disease patients and evaluate either only self-efficacy or only self-management. The aim of this study was to adapt the Heart Health Self-efficacy and Self-Management Scale (HH-SESM) into Turkish and to investigate its validity and reliability in patients with coronary heart disease. The study is conducted in Cardiology outpatient clinics of Karaman Training and Research Hospital. Before the study, the purpose and content of the study will be explained to the participants and an informed consent form will be obtained from the participants. Since the sample size in validity and reliability studies should be at least 10 times the total number of scale items, at least 120 individuals will be included in the study as the number of items x number of options (12 x 10 = 120). Detailed medical history and sociodemographic information (age, gender, height, weight, body mass index, disease duration (months), occupation, daily working hours, educational status, sports/exercise habits) will be recorded. In order to measure self-management and self-efficacy levels, patients will be administered the HH-SESM, Self-care management in chronic diseases scale- Self-care subgroup questions and General self-efficacy scales.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with coronary heart disease for at least 6 months
* Speaking Turkish
* to be able to read and write
* Being over 18 years old
* volunteering to participate in the study

Exclusion Criteria:

* Having a serious psychiatric illness such as panic disorder or major depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer who had been diagnosed coronary heart disease for at least 6 months
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
validity and reliability of Turkish Heart Health Self-efficacy and Self-Management Scale | within 24 hours of admission
  It will be applied to the patients as a questionnaire in order to make the Turkish validity and reliability of the Heart Health Self-efficacy and Self-Management Scale. Scores ≥36 can be interpreted as high self-efficacy and high self-management. The scale consists of 12 items and is scored using a 4-point Likert system. But since there is also an invalid answer option, people can get a minimum score of 0 and a maximum score of 48. Scores ≥36 can be interpreted as high self-efficacy and high self-management. Scores between 24 - 35 can be interpreted as adequate self-efficacy and adequate self-management. Scores ≤24 can be interpreted as low self-efficacy and low self-management.

SECONDARY OUTCOMES:
Self-Care Management Scale in chronic diseases | within 24 hours of admission
  For the external construct validity statistical method, the self-management level of the individuals will be determined with the Self-Care Management in Chronic Diseases Scale, which has been previously validated and reliable in Turkish. The scale consists of 20 items. The scale is analysed over the total score. 5-point Likert system is used in scoring, with 1 point for strongly disagree and 5 points for strongly agree.
  Individuals can get a maximum score of 100 and a minimum score of 20. A high score indicates high general self-efficacy; a low score indicates low self-efficacy.
General self-efficacy scale | within 24 hours of admission
  For the external construct validity statistical method, the self-efficacy level of the individuals will be determined with the general self-efficacy scale, which has been previously validated and reliable in Turkish. The scale consists of 10 items. The scale is analysed over the total score. Points are given to the items according to the answers.
  Completely wrong = 1 point Somewhat correct = 2 points Moderately correct = 3 points Completely correct = 4 points
  Individuals can get a maximum score of 40 and a minimum score of 10. A high score indicates high general self-efficacy; a low score indicates low self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoğlu Mehmetbey University, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Tunc Suygun E, Vardar Yagli N, Suygun H, Saglam M. Validity and reliability of the Turkish translation of the heart health self-efficacy and self-management scale in patients with chronic heart disease. BMC Psychol. 2025 Nov 3;13(1):1210. doi: 10.1186/s40359-025-03539-6. PMID 41185050